CLINICAL TRIAL: NCT01354561
Title: Effect of Airway Clearance Therapy on the Cardiac Autonomic Modulation in Hospitalized Paediatric Patients
Brief Title: Respiratory Physical Therapy on the Cardiac Autonomic Modulation Paediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Hugo C.D. Souza, Ph.D., University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USP10
Record Dates: First submitted 2011-05-09; First posted 2011-05-17 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Viral Bronchiolitis
Keywords: respiratory physiotherapy; cardiac autonomic modulation; paediatric patients
MeSH Terms: conditions — Bronchiolitis, Viral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Sham Comparator): Physiotherapy in the control group were also done at hospital, in dorsal decubitus position at 30-degree elevation, all receiving the same treatment given for the paediatric inpatients, except nasotracheal suction, which was not performed due to ethical reasons.
  Interventions: Procedure: Respiratory physical therapy
- respiratory disease group (Active Comparator): Respiratory disease group consisting of hospitalized children with acute viral bronchiolitis
  Interventions: Procedure: Respiratory physical therapy

INTERVENTIONS:
Procedure: Respiratory physical therapy — Respiratory physical therapy using airway clearance techniques was conducted by a physiotherapist according to a detailed clinical evaluation of each patient, consisting of thoracic percussion, manual vibration, postural drainage, and cough stimulation.
  Other Names: chest therapy

SUMMARY:
The present study investigated the influence of respiratory affections on the heart rate variability (HRV) of paediatric patients. We have hypothesised that respiratory physiotherapy would promote a beneficial effect on the cardiac autonomic modulation. Twenty-four children, who were divided into respiratory disease group (RG) and control (CG) groups, were studied. Analysis of HRV was performed with the RG in the dorsal decubitus position during four different moments: basal record (30 minutes); 5 minutes after respiratory physiotherapy by means of airway clearance techniques (10-minute record); 5 minutes after nasotracheal suction (10-minute record); and 40 minutes after nasotracheal suction (30-minute record). CG group was submitted to the same protocol, except nasotracheal suction, which was not performed due to ethical reasons.

DETAILED DESCRIPTION:
The study of heart rate variability (HRV) is a method allowing non-invasive and selective evaluation of the changes in cardiac autonomic modulation. Its use in several clinical situations has provided important information, serving as an evaluation instrument for a better understanding of the involvement of the autonomic nervous system in various physiopathological situations.

With regard to the applicability of HRV analysis in paediatric populations, it is known that the maturity progression of sympathetic and vagal divisions is accompanied by a growing increase in autonomic modulation over the pre- and post-natal periods. In turn, a few studies have addressed the association between pathological paediatric conditions and changes in the cardiac autonomic modulation, consequently, HRV.

Among these pathologies, the respiratory affections are the main factors of morbidity and mortality in children, since newborns have peculiar aspects involving the respiratory system that can easily lead to a lung failure. Within this context, one can note the importance of the respiratory physiotherapy as an intervention using specific procedures in each case in order to decrease the airway resistance and improve the ventilation/perfusion ratio, thus improving the respiratory function and minimising the clinical severity. Consequently, in patients suffering from obstructive pathologies or neuromuscular dysfunctions, which makes cough an inefficient mechanism, physiotherapy can help them to recover from their condition.

Therefore, the respiratory physiotherapy has influence on the several hospitalisation phases, contributing to make the hospital stays shorter and less difficult to the paediatric inpatient and promoting a more humanised and more efficient environment based on the patient's needs. In this sense, it is possible that the paediatric inpatients present important alterations in their cardiovascular autonomic control, since constant oscillations in the cardiac and hemodynamic parameters are observed. However, studies correlating HRV with respiratory pathological conditions in paediatric inpatients are rare, either before or after the respiratory physiotherapy procedures, such as application of airway clearance techniques.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized children

Exclusion Criteria:

* age above 12 months;
* presence of cardiovascular disease or chronic respiratory disease;
* prescription of vasoactive drugs or sedatives;
* invasive mechanical ventilation;
* children on contact or respiratory isolation.

Ages: 2 Months to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2007-02; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | basal record
  The heart rate (HR) was recorded with the children in the dorsal decubitus position at 30-degree elevation during 30 minutes before performing the respiratory physiotherapy using airway clearance techniques (ACTs)

SECONDARY OUTCOMES:
Heart Rate Variability | 5 minutes after ACTs
  The heart rate (HR) was recorded with the children in the dorsal decubitus position at 30-degree elevation during 10 minutes after 5 minutes performing the respiratory physiotherapy using airway clearance techniques(ACTs)
Heart Rate Variability | 5 minutes after nasotracheal suction
  The heart rate (HR) was recorded with the children in the dorsal decubitus position at 30-degree elevation after 5 minutes nasotracheal suction (10-minutes record).
Heart Rate Variability | 40 minutes after nasotracheal suction
  The heart rate (HR) was recorded with the children in the dorsal decubitus position at 30-degree elevation during 40 minutes after nasotracheal suction (30-minute record).

CONTACTS AND LOCATIONS:
Overall Officials: Hugo CD Souza, Ph.D., Study Director — University of Sao Paulo
Locations (1):
- University of São Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Sant'Ana JE, Pereira MG, Dias da Silva VJ, Dambros C, Costa-Neto CM, Souza HC. Effect of the duration of daily aerobic physical training on cardiac autonomic adaptations. Auton Neurosci. 2011 Jan 20;159(1-2):32-7. doi: 10.1016/j.autneu.2010.07.006. Epub 2010 Aug 13. PMID 20708981
- [Derived] Jacinto CP, Gastaldi AC, Aguiar DY, Maida KD, Souza HC. Physical therapy for airway clearance improves cardiac autonomic modulation in children with acute bronchiolitis. Braz J Phys Ther. 2013 Nov-Dec;17(6):533-40. doi: 10.1590/S1413-35552012005000120. Epub 2013 Nov 1. PMID 24271093
- See also: Related Info — http://www.fmrp.usp.br